CLINICAL TRIAL: NCT03497403
Title: Socket Preservation Revisited: RCT to Study the Three-dimensional Changes of Hard and Soft Tissue Comparing Two Distinct Surgical Protocols
Brief Title: Socket Preservation Procedure Studying Soft and Hard Tissue Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Dental Medicine (Other)
Collaborators: Valeant Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Heather Hong, Principle Investigator, Harvard School of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-3772
Record Dates: First submitted 2018-04-05; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Ridge Preservation; Bone Regeneration

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of two groups in parallel for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Socket preservation control. After tooth extraction, bone graft is applied to socket and a non-cross-linked membrane is used in primary intentional healing.
  Interventions: Procedure: Socket preservation control
- Experimental (Experimental): Socket preservation experimental. After tooth extraction, bone graft is applied to socket and a cross-linked membrane is used in secondary intention healing.
  Interventions: Procedure: Socket preservation experimental

INTERVENTIONS:
Procedure: Socket preservation control — After a tooth was extracted, the adjacent gum tissue was fully reflected, bone graft (FDBA) and non-cross-linked barrier membrane (Bio-Gide) were applied to the defect. The site was stabilized with sutures. Patients were followed for 6 months post operatively.
  Arms: Control
Procedure: Socket preservation experimental — After a tooth was extracted, the adjacent gum tissue was minimally reflected, bone graft (FDBA) and cross-linked barrier membrane (OssixPlus) were applied to the defect. The site was stabilized with sutures. Patients were followed for 6 months post operatively.
  Arms: Experimental

SUMMARY:
Two different surgical protocols for socket preservation were compared. Soft and hard tissue outcomes were measured clinically and radiographically at baseline and six months post operatively.

DETAILED DESCRIPTION:
The effect of different surgical techniques for socket preservation on soft tissue parameters has seldom been investigated. The aim of this study was to evaluate One with a cross-linked membrane used in secondary intention healing and the other with a non-cross-linked membrane used in primary intentional healing. Thirty subjects requiring tooth extraction were randomly allocated to either control group C (allograft covered with a non-cross-linked collagen membrane with primary closure) or experimental group E (allograft covered with cross-linked collagen membrane left exposed). Sites were surgically re-entered at 6-months. Soft and hard tissue measurements, cone beam computed tomography (CBCT) and cast measurements were taken at baseline & 6-months.

ELIGIBILITY:
Inclusion Criteria:

1. between 20-80 years of age
2. healthy with no conditions that could alter wound healing
3. requiring the extraction of a non-molar tooth with two neighboring teeth on either side and intact bony walls
4. a tooth requiring extraction that is treatment planned for implant placement
5. willing to participate in the study and sign the informed consent
6. willing to receive clinical exams, radiographs, surgery, two and six week post-operative exams and six month re-entry exam.

Exclusion Criteria:

1. systemic conditions which could alter wound healing
2. tooth anatomy requiring aggressive bone removal or greater flap reflection for extraction
3. severe local infection at extraction site
4. a tooth exhibiting severe resorption of buccal or lingual plates
5. absence of keratinized tissue buccal to the tooth to be extracted
6. severely reduced vestibular depth (≤ 3.0 mm) at the tooth to be extracted.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Keratinized tissue width | 6 months
  Keratinized gingival tissue width measured from the free gingival margin to the muco-gingival junction.

SECONDARY OUTCOMES:
Keratinized tissue thickness | 6 months
  Keratinized gingival tissue thickness measured with a needle and stopper 3mm from the free gingival margin.
Vestibular Depth | 6 months
  The distance from the free gingival margin to the apical extent of the vestibule measured with a probe.
CEJ-FGM | 6 months
  The distance from the tooth's cervical enamel junction (CEJ) to the free gingival margin (FGM) was taken with a probe.
Ridge Width | 6 months
  After the gum tissue is reflected, the width of the ridge 6mm from the crest was measured with a caliper.
CEJ- Buccal crest | 6 months
  The distance from the tooth's cervical enamel junction and the top of the buccal bone crest was taken with a probe.
CBCT bone height | 6 months
  CBCT scans were taken and the alveolar ridge height was then measured.
CBCT bone width | 6 months
  CBCT scans were taken and the alveolar ridge width was then measured.
Cast ridge width | 6 months
  Dental impressions were taken and stone casts obtained from them.The ridge width was then measured with calipers.
Cast ridge volume | 6 months
  Dental impressions were taken and stone casts obtained from them.The ridge volume was measured using an optical scanner.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Machtei, DMD, Principal Investigator — Harvard School of Dental Med.
Locations (1):
- Harvard School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT03497403/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-05-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT03497403/Prot_SAP_001.pdf